CLINICAL TRIAL: NCT02088541
Title: A Randomized, Open Label, Phase 2 Study of the Selective Inhibitor of Nuclear Export (SINE) Selinexor (KPT-330) Versus Specified Physician's Choice in Patients ≥ 60 Years Old With Relapsed or Refractory Acute Myeloid Leukemia (AML) Who Are Ineligible for Intensive Chemotherapy and/or Transplantation
Brief Title: Selinexor (KPT-330) in Older Patients With Relapsed AML
Acronym: SOPRA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Karyopharm Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KCP-330-008
Record Dates: First submitted 2014-03-09; First posted 2014-03-17 (Estimated); Results first posted 2020-10-08 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Acute Myeloid Leukemia (AML)
Keywords: Relapsed/Refractory Acute Myeloid Leukemia; Acute Myeloid Leukemia; AML; Karyopharm; Selinexor; KPT-330
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — selinexor; Hydroxyurea; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Selinexor approximately 55 mg/m^2 (60 to 120 mg based on BSA) (Experimental): Participants under protocol versions (PV) less than (<) 5.0 (those who had one prior line of acute myeloid leukemia (AML) therapy), receive oral selinexor tablets at a dose of approximately 55 mg/m^2 (milligrams per square meter) (60 to 120 mg based on body surface area [BSA]) twice weekly, on Day 1 and 3 of each week of 4-week cycle (28 days per cycle).
  Interventions: Drug: Selinexor
- Selinexor 60 mg (PV <5) (Equivalent to 35 mg/m^2) (Experimental): Participants under PV < 5.0 (those who had one prior line of AML therapy), receive oral selinexor tablets at a fixed dose of 60 mg (equivalent to 35 mg/m^2), based on BSA, twice weekly, on Day 1 and 3 of each week of 4-week cycle (28 days per cycle).
  Interventions: Drug: Selinexor
- Selinexor 60 mg (PV >=5) (Equivalent to 35 mg/m^2) (Experimental): Participants under PV >= 5 (PV 5: those who had at least one prior line of AML therapy, PV 5.1: who had at least two prior line of AML therapy), receive oral selinexor tablets at a dose of 60 mg (equivalent to 35 mg/m^2) twice weekly, on Day 1 and 3 of each week of 4-week cycle (28 days per cycle).
  Interventions: Drug: Selinexor
- Physician's Choice 1 (PV <5) (Active Comparator): Participants under PV < 5.0 (those who had one prior line of AML therapy) received Best Supportive Care (BSC) which included blood product transfusions, antimicrobials, growth factors as needed, and hydroxyurea.
  Interventions: Drug: Hydroxyurea
- Physician's Choice 2 (PV >=5) (Active Comparator): Participants under PV >= 5 (PV 5: those who had at least one prior line of AML therapy, PV 5.1: who had at least two prior line of AML therapy), received BSC along with subcutaneous injection of arabinoside cytosine (Ara-C), 20 mg, twice daily, for 10 days, repeated at 28 to 42 day intervals.
  Interventions: Drug: Ara-C

INTERVENTIONS:
Drug: Selinexor — Selinexor oral tablet.
  Other Names: KPT-330
  Arms: Selinexor 60 mg (PV <5) (Equivalent to 35 mg/m^2); Selinexor 60 mg (PV >=5) (Equivalent to 35 mg/m^2); Selinexor approximately 55 mg/m^2 (60 to 120 mg based on BSA)
Drug: Hydroxyurea
  Other Names: Hydroxycarbamide
  Arms: Physician's Choice 1 (PV <5)
Drug: Ara-C — Ara-C Subcutaneous Injection.
  Other Names: Cytarabine; Cytosine arabinoside; Cytosar-U; Depocyt
  Arms: Physician's Choice 2 (PV >=5)

SUMMARY:
This is a randomized, multicenter, open-label, phase 2 study of the SINE compound, selinexor given orally versus specified investigator choices (one of three potential salvage therapies). Participants age ≥ 60 years with relapsed or refractory AML of any type except for AML M3, after one prior therapy only, who have never undergone and who are not currently eligible for stem cell transplantation and are currently deemed unfit for intensive chemotherapy.

DETAILED DESCRIPTION:
This is a randomized, multicenter, open-label phase 2 study of the SINE compound, selinexor given orally versus restricted investigator choice (i.e., one of three potential salvage therapies).

Participants who have never been transplant eligible, are currently deemed unfit for intensive chemotherapy, ≥ 60 years old, who have AML (except Acute Promyelocytic Leukemia: APL, AML M3) after one prior treatment of either hypomethylating agent or a regimen including Ara-C, and are meeting the inclusion and exclusion criteria will be randomized to receive either oral selinexor or physician's choice (one of three potential treatments: best supportive care (BSC) alone, or BSC + hypomethylating agent, or BSC + low dose Ara-C until disease progression, death or intolerance has occurred.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 years with relapsed or refractory AML of any type except for acute promyelocytic leukemia (APL; AML M3), after at least 1 prior AML therapy , who have never undergone, and who are not currently eligible for, stem cell transplantation, and are currently deemed unfit for intensive chemotherapy.
* Eastern Cooperative Oncology Group (ECOG) ≤ 2.
* Must have available archival or recently acquired bone marrow biopsy/aspiration or tumor tissue for central review to be eligible.
* Relapsed or refractory AML, defined as either: recurrence of disease after a complete remission (CR), or failure to achieve CR with initial therapy.
* Must have received at least 1 prior line of AML therapy given at standard doses and must have progressed after their most recent therapy. Prior therapy must have included: a hypomethylating agent with at least 2 cycles.
* At least 2 weeks must have elapsed since the last anti-leukemia treatment (with the exception of hydroxyurea) before first dose in this study.

Exclusion Criteria:

* Treatment with any investigational agent within 3 weeks prior to first dose in this study.
* Presence of central nervous system (CNS) leukemia.
* In blast transformation of chronic myeloid leukemia (CML). Prior myelodysplastic syndrome (MDS) is acceptable; prior treatment for MDS does not count as an AML therapy.
* Major surgery within 2 weeks of first dose of study drug. Participants must have recovered from the effects of any surgery performed greater than 2 weeks previously.
* Concurrent active malignancy under treatment.
* Known active hepatitis B virus (HBV) or C virus (HCV) infection; or known to be positive for HCV ribonucleic acid (RNA) or HBsAg (HBV surface antigen).
* Known HIV infection.
* Unable to swallow tablets, or participants with malabsorption syndrome, or any other disease significantly affecting gastrointestinal function.
* Participants whose AML is classified as favorable according to the European LeukemiaNet (ELN) disease risk assessment.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 317 (Actual)
Dates: Start 2014-03; Primary Completion 2018-01-08 (Actual); Study Completion 2018-01-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (78):
- United States (26):
  - Jonsson Comprehensive Cancer Center / University of California, Los Angeles, Los Angeles, California
  - Sutter Oncology & Hematology, Sacramento, California
  - Stanford Cancer Institute / Stanford University, Stanford, California
  - Colorado Blood Cancer Institute/Sarah Cannon Research Institute, Denver, Colorado
  - Yale Cancer Center / Yale University, New Haven, Connecticut
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Winship Cancer Institute / Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Chicago Medicine, Chicago, Illinois
  - University of Kansas Hospital, Kansas City, Kansas
  - Sidney Kimmel Comprehensive Cancer Center / John Hopkins University, Baltimore, Maryland
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Westchester Medical Center / New York Medical College, Hawthorne, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - New York Presbyterian Hospital / Weill Cornell Medical College, New York, New York
  - Duke Cancer Care, Durham, North Carolina
  - Gabrail Cancer Center, Canton, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Milton S. Hershey Medical Center / Penn State, Hershey, Pennsylvania
  - Tennessee Oncology/Sarah Cannon Research Institute, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center / Vanderbilt University, Nashville, Tennessee
  - MD Anderson Cancer Center / University of Texas, Houston, Texas
  - Texas Transplant Institute/Sarah Cannon Research Institute, San Antonio, Texas
- Canada (3):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - Sir Mortimer B. Davis Jewish General Hospital / McGill University, Montreal, Quebec
- Denmark (4):
  - Aarhus University Hospital, Aarhus
  - Department of Haematology, National University Hospital, Rigshospitalet, Copenhagen
  - Herlev Hospital, Herlev
  - Odense University Hospital, Department of Hematology, Odense
- France (5):
  - CHU Bordeaux- Hôpital Haut Lévêque, Bordeaux
  - Centre Hospitalier Lyon, Lyon
  - Hopital Saint Louis, Paris
  - Hôpital Avicenne, Paris
  - Institut Universitaire du Cancer Toulouse, Toulouse
- Germany (8):
  - Stellvertretende Klinikleiterin Charité, Campus Benjamin Franklin, Berlin
  - Ev. Diakonie-Krankenhaus Gemeinnutzige GMBH Medizinische Klinik 2, Bremen
  - UNIVERSITÄTSKLINIKUM TU DRESDEN Medizinische Klinik und Poliklinik I,, Dresden
  - University Hospital Frankfurt, Frankfurt
  - Medizinische Hochschule Hannover (Hannover Medical School) Dept. of Hematology, Hemostasis, Oncology, and Stem Cell Transplantation, Hanover
  - Abteilung Hämatologie, internistische Onkologie und Hämostaseologie, Leipzig
  - UNIVERSITY HOSPITAL OF MÜNSTER Medizinische Klinik und Poliklinik A, Universitätsklinikum Münster, Münster
  - Universitätsklinikum Ulm, Ulm
- Israel (7):
  - Sororka MC, Beersheba
  - Rambam Health Care Campus, Haifa
  - Wolfson Medical Center, Holon
  - Hadassah Medical Center, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Tel Aviv Sourasky Medical Centre, Tel Aviv
  - Chaim Sheba Medical Center, Tel Litwinsky
- Italy (3):
  - AOU Ospedali Riuniti di Ancona, Ancona
  - A.O Spedali Civili di Brescia, Brescia
  - AORN Cardarelli / UOSC di Ematologia con TMO, Naples
- Netherlands (7):
  - AMC, Academisch Medisch Centrum Afdeling Klinische Hematologie, Amsterdam
  - VU University Medical Center, Amsterdam
  - Universitair Medisch Centrum Groningen Department of Haematology, Groningen
  - Radboud University Medical Center Department of Haematology (476), Nijmegen
  - Erasmus MC, location Daniel den Hoed, Rotterdam
  - University Medical Center Utrecht, Utrecht
  - Isala Kliniecken Zwolle, Zwolle
- Poland (4):
  - Wojewódzki Szpital Specjalistyczny im. M. Kopernika, Klinika Hematologii, Lodz
  - Samodzielny Publiczny Zakład Opieki Zdrowotnej Ministerstwa Spraw Wewnętrznych, Olsztyn
  - Instytut Hematologii i Transfuzjologii, Warsaw
  - Samodzielny Publiczny Szpital Kliniczny Nr 1 we Wrocławiu, Wroclaw
- Spain (4):
  - ICO Badalona, Badalona
  - Hospital del Mar, Barcelona
  - Hospital Universitario de Salamanca Servicio de Hematologia, Salamanca
  - Hospital Universitario y Politécnico La Fe, Valencia
- United Kingdom (7):
  - Northwick Park Hospital, Harrow, England
  - Royal Liverpool University Hospital, Dept of Cellular and Molecular Physiology, Molecular and Clinical Cancer Medicine, Liverpool, Lancashire
  - Royal Marsden NHS Trust, Sutton, Surrey
  - University Hospital Wales, Cardiff, Wales
  - Hull and East Yorkshire Hospitals NHS Trust Queens Centre for Oncology and Haematology, Hull, Yorkshire
  - Ninewells Hospital and Medical School NHS Tayside, Dundee
  - Plymouth Hospitals NHS Trust/Derriford Hospital, Plymouth

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Sweet K, Bhatnagar B, Dohner H, Donnellan W, Frankfurt O, Heuser M, Kota V, Liu H, Raffoux E, Roboz GJ, Rollig C, Showel MM, Strickland SA Jr, Vives S, Tang S, Unger TJ, Joshi A, Shen Y, Alvarez MJ, Califano A, Crochiere M, Landesman Y, Kauffman M, Shah J, Shacham S, Savona MR, Montesinos P. A 2:1 randomized, open-label, phase II study of selinexor vs. physician's choice in older patients with relapsed or refractory acute myeloid leukemia. Leuk Lymphoma. 2021 Dec;62(13):3192-3203. doi: 10.1080/10428194.2021.1950706. Epub 2021 Jul 29. PMID 34323164

RESULTS

PARTICIPANT FLOW:
Groups:
- Selinexor Approximately 55 mg/m^2 (60 to 120 mg Based on BSA): Participants under protocol versions (PV) less than (<) 5.0 (those who had one prior line of acute myeloid leukemia (AML) therapy), received oral selinexor tablets at a dose of approximately 55 mg/m^2 (milligrams per square meter) (60 to 120 mg based on body surface area [BSA]) twice weekly, on Day 1 and 3 of each week of 4-week cycle (28 days per cycle).
- Selinexor 60 mg (PV <5) (Equivalent to 35 mg/m^2): Participants under PV < 5.0 (those who had one prior line of AML therapy), received oral selinexor tablets at a fixed dose of 60 mg (equivalent to 35 mg/m^2), twice weekly, on Day 1 and 3 of each week of 4-week cycle (28 days per cycle).
- Selinexor 60 mg (PV >=5) (Equivalent to 35 mg/m^2): Participants under PV greater than or equal to (>=) 5 (PV 5: those who had at least one prior line of AML therapy, PV 5.1: who had at least two prior line of AML therapy), received oral selinexor tablets at a dose of 60 mg (equivalent to 35 mg/m^2) twice weekly, on Day 1 and 3 of each week of 4-week cycle (28 days per cycle).
- Physician's Choice 2 (PV >=5): Participants under PV>= 5 (PV 5: those who had at least one prior line of AML therapy, PV 5.1: who had at least two prior line of AML therapy), received BSC along with subcutaneous injection of arabinoside cytosine (Ara-C), 20 mg, twice daily, for 10 days, repeated at 28 to 42 day intervals.
Period: Overall Study
Arm/Group | Selinexor Approximately 55 mg/m^2 (60 to 120 mg Based on BSA) | Selinexor 60 mg (PV <5) (Equivalent to 35 mg/m^2) | Selinexor 60 mg (PV >=5) (Equivalent to 35 mg/m^2) | Physician's Choice 1 (PV <5) | Physician's Choice 2 (PV >=5)
Started | 71 | 27 | 117 | 44 | 58
Safety Population | 71 | 27 | 115 | 39 | 45
Intent-to-treat (ITT) Population | 0 | 0 | 118 (1 randomized to Selinexor 60mg (PV>=5) but treated with physician choice 2, counted under this arm.) | 0 | 57
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 71 | 27 | 117 | 44 | 58
Not completed — Adverse Event | 3 | 0 | 3 | 3 | 0
Not completed — Death | 51 | 21 | 85 | 28 | 38
Not completed — Lost to Follow-up | 2 | 0 | 1 | 0 | 0
Not completed — Physician Decision | 2 | 1 | 2 | 0 | 2
Not completed — Disease progression | 7 | 1 | 2 | 3 | 1
Not completed — Study terminated by sponsor | 1 | 1 | 12 | 2 | 6
Not completed — Withdrawal by Subject | 3 | 2 | 9 | 7 | 10
Not completed — Other | 2 | 1 | 3 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety Population included all participants who received any amount of study treatment and was the primary population for the analysis of safety outcome measure.
Groups:
- Selinexor Approximately 55 mg/m^2 (60 to 120 mg Based on BSA): Participants under PV < 5.0 (those who had one prior line of AML therapy), received oral selinexor tablets at a dose of approximately 55 mg/m^2 (60 to 120 mg based on BSA) twice weekly, on Day 1 and 3 of each week of 4-week cycle (28 days per cycle).
- Selinexor 60 mg (PV<5) (Equivalent to 35 mg/m^2): Participants under PV < 5.0 (those who had one prior line of AML therapy), received oral selinexor tablets at a fixed dose of 60 mg (equivalent to 35 mg/m^2), based on BSA, twice weekly, on Day 1 and 3 of each week of 4-week cycle (28 days per cycle).
- Selinexor 60 mg (PV >=5) (Equivalent to 35 mg/m^2): Participants under PV >= 5 (PV 5: those who had at least one prior line of AML therapy, PV 5.1: who had at least two prior line of AML therapy), received oral selinexor tablets at a dose of 60 mg (equivalent to 35 mg/m^2) twice weekly, on Day 1 and 3 of each week of 4-week cycle (28 days per cycle).
- Total: Total of all reporting groups
Arm/Group | Selinexor Approximately 55 mg/m^2 (60 to 120 mg Based on BSA) | Selinexor 60 mg (PV<5) (Equivalent to 35 mg/m^2) | Selinexor 60 mg (PV >=5) (Equivalent to 35 mg/m^2) | Physician's Choice 1 (PV <5) | Physician's Choice 2 (PV >=5) | Total
Number analyzed (Participants) | 71 | 27 | 115 | 39 | 45 | 297
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.4 (6.49) | 73.2 (4.64) | 73.6 (5.99) | 72.6 (5.24) | 74.2 (5.92) | 73.2 (5.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 11 | 46 | 17 | 15 | 115
  Male | 45 | 16 | 69 | 22 | 30 | 182
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 9 | 4 | 6 | 26
  Not Hispanic or Latino | 65 | 23 | 93 | 34 | 31 | 246
  Unknown or Not Reported | 2 | 1 | 13 | 1 | 8 | 25
Race/Ethnicity, Customized [Number; unit: Count of Participants]
  White | 67 | 22 | 95 | 39 | 37 | 260
  Black or African American | 3 | 1 | 3 | 0 | 0 | 7
  Asian | 0 | 2 | 0 | 0 | 0 | 2
  Other | 0 | 1 | 15 | 0 | 6 | 22
  Unknown | 1 | 1 | 2 | 0 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival was defined as the time (in days) from the date of randomization to the date of death due to any cause. Participants last known to be alive were censored at date of last contact.
Time Frame: Baseline until disease progression or discontinuation from the study, or death, whichever occurred first (up to a maximum of approximately 104 weeks)
Population: Intent-to-treat (ITT) population included all participants who were randomized to study treatment under PV>=5.0, regardless of whether or not they received study treatment. One participant was randomized to receive selinexor 60 mg (PV>=5) but was treated with physician's choice 2. Hence, this participant was counted under selinexor 60 mg (PV>=5).
Measure: Median (95% Confidence Interval); unit: Days
Groups:
- Selinexor 60 mg (PV >=5) (Equivalent to 35 mg/m^2): Participants under PV >=5 (PV 5: those who had at least one prior line of AML therapy, PV 5.1: who had at least two prior line of AML therapy), received oral selinexor tablets at a dose of 60 mg (equivalent to 35 mg/m^2) twice weekly, on Day 1 and 3 of each week of 4- week cycle (28 days per cycle).
Arm/Group | Selinexor 60 mg (PV >=5) (Equivalent to 35 mg/m^2) | Physician's Choice 2 (PV >=5)
Number analyzed (Participants) | 118 | 57
Days | 94.0 [78.0 to 158.0] | 170.0 [111.0 to 220.0]
Statistical Analysis 1: Comparison: Selinexor 60 mg (PV >=5) (Equivalent to 35 mg/m^2) vs Physician's Choice 2 (PV >=5); Test type: Superiority; p = 0.4221, Log Rank; Hazard Ratio (HR) = 1.18, 95% CI 2-sided [0.79 to 1.75]

2. Secondary Outcome: Percentage of Participants With Overall Survival of at Least 3 Months (OS3.0)
Description: Overall survival was defined as the time (in days) from the date of randomization to the date of death due to any cause. Participants last known to be alive were censored at date of last contact. Analysis was performed using Kaplan-Meier method.
Time Frame: From randomization (Day 1) up to 3 months
Population: ITT population included all participants who were randomized to study treatment under PV >=5.0, regardless of whether or not they received study treatment. One participant was randomized to receive selinexor 60 mg (PV>=5) but was treated with physician's choice 2. Hence, this participant was counted under selinexor 60 mg (PV>=5).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Selinexor 60 mg (PV >=5) (Equivalent to 35 mg/m^2) | Physician's Choice 2 (PV >=5)
Number analyzed (Participants) | 118 | 57
Percentage of participants | 53.49 [43.54 to 62.44] | 70.73 [55.60 to 81.52]
Statistical Analysis 1: Comparison: Selinexor 60 mg (PV >=5) (Equivalent to 35 mg/m^2) vs Physician's Choice 2 (PV >=5); Test type: Superiority; p = 0.9464, Log Rank

3. Secondary Outcome: Percentage of Participants With Complete Remission Rate (CRR) for Those Who Achieved Complete Remission (CR)
Description: CRR was analyzed using International Working Group (IWG) 2003 criteria, as the difference in the proportions of participants with IWG results of CR. CR per IWG 2003 criteria was defined as morphologic presence of < 5 percentage (%) myeloblasts in bone marrow, the absence of circulating blasts, hematologic recovery (as evidenced by a peripheral blood absolute neutrophil count (ANC) > 1000 cells/microliter (microL) and platelet count > 100,000/microL, with no need for red blood cell (RBC) transfusions), and the absence of extramedullary disease.
Time Frame: as for outcome 1
Population: ITT population included all participants who were randomized to study treatment under PV>=5.0, regardless of whether or not they received study treatment. One participant was randomized to receive selinexor 60 mg (PV>=5) but was treated with physician's choice 2. Hence, this participant was counted under selinexor 60 mg (PV>=5).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Selinexor 60 mg (PV >=5) (Equivalent to 35 mg/m^2) | Physician's Choice 2 (PV >=5)
Number analyzed (Participants) | 118 | 57
Percentage of participants | 5.1 [1.9 to 10.7] | 0 [0.0 to 6.3]
Statistical Analysis 1: Comparison: Selinexor 60 mg (PV >=5) (Equivalent to 35 mg/m^2) vs Physician's Choice 2 (PV >=5); Test type: Superiority; p = 0.0986, Cochran-Mantel-Haenszel

4. Secondary Outcome: Median Disease-Free Survival (DFS) for Participants Who Achieved Complete Remission (CR)
Description: DFS for CRR based on IWG criteria, was calculated from the first date of response of CR to the date of progression or recurrence, or date of death if progression or recurrence did not occur. Participants who discontinued prior to disease progression or recurrence or did not progress as of the time of the analysis were censored at the time of last radiologic assessment. CR per IWG 2003 criteria was defined as morphologic presence of < 5 % myeloblasts in bone marrow, the absence of circulating blasts, hematologic recovery (as evidenced by a peripheral blood ANC > 1000 cells/microL and platelet count > 100,000/microL, with no need for RBC transfusions), and the absence of extramedullary disease.
Time Frame: as for outcome 1
Population: ITT population:all participants who randomized to study treatment under PV>=5.0, regardless of whether or not they received study treatment. This outcome measure(OM) was only defined for CR participants. For Physician Choice 2,there was zero CR participants."Overall Number of Participants Analyzed (N)": Number of participants evaluable for this OM.
Measure: Median (95% Confidence Interval); unit: Days
Groups:
- Selinexor 60 mg (PV >=5) (Equivalent to 35 mg/m^2): Participants under PV >=5, received oral selinexor tablets at a dose of 60 mg (equivalent to 35 mg/m^2) twice weekly, on Day 1 and 3 of each week of 4-week cycle (28 days per cycle).
Arm/Group | Selinexor 60 mg (PV >=5) (Equivalent to 35 mg/m^2) | Physician's Choice 2 (PV >=5)
Number analyzed (Participants) | 6 | 0
Days | 121.0 [49.0 to NA] — Upper limits of 95% confidence Interval (CI) was not estimable due to less number of participants and events. |

5. Secondary Outcome: Percentage of Participants With Modified Complete Remission Rate (mCRR) for Those Who Achieved Complete Remission (CR) or Complete Remission With Incomplete Hematologic Recovery (Cri)
Description: mCRR was defined as the point estimate of the percentage of participants who had CR, CRi, or CRp. Responses defined as per IWG 2003 response criteria: Morphologic CR:< 5% myeloblasts in bone marrow, the absence of circulating blasts, hematologic recovery (as evidenced by a peripheral blood ANC > 1000 cells/microL and platelet count > 100,000/microL, with no need for RBC transfusions), and the absence of extramedullary disease. Morphologic CRp: All criteria for CR except for residual neutropenia (<1x10^9/L) or thrombocytopenia (<100 x10^9/L), Cri (< 5% bone marrow blasts with residual neutropenia [ANC < 1000 cells/microL] or thrombocytopenia [platelets < 100,000/microL]), normal maturation of all cellular components in the bone marrow, no extramedullary disease and transfusion independent.
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Selinexor 60 mg (PV >=5) (Equivalent to 35 mg/m^2) | Physician's Choice 2 (PV >=5)
Number analyzed (Participants) | 118 | 57
Percentage of participants | 11.9 [6.6 to 19.1] | 3.5 [0.4 to 12.1]
Statistical Analysis 1: Comparison: Selinexor 60 mg (PV >=5) (Equivalent to 35 mg/m^2) vs Physician's Choice 2 (PV >=5); Test type: Superiority; p = 0.0844, Cochran-Mantel-Haenszel

6. Secondary Outcome: Median Disease-Free Survival (DFS) for Participants Who Achieved Complete Remission or CR With Incomplete Hematologic Recovery (CRi) or Complete Remission With Incomplete Platelet Recovery (CRp)
Description: DFS based on IWG criteria was defined as the duration from start of the complete response achieved until disease progression or death from any cause. Responses defined by IWG 2003 Response Criteria: Morphologic CR: < 5% myeloblasts in bone marrow, the absence of circulating blasts, hematologic recovery (as evidenced by a peripheral blood ANC > 1000 cells/microL and platelet count > 100,000/microL, with no need for RBC transfusions), and the absence of extramedullary disease. Morphologic CRp: All criteria for CR except for residual neutropenia (<1x10^9/L) or thrombocytopenia (<100 x10^9/L), Cri (< 5% bone marrow blasts with residual neutropenia [ANC < 1000 cells/microL] or thrombocytopenia [platelets < 100,000/microL]), normal maturation of all cellular components in the bone marrow, no extramedullary disease and transfusion independent.
Time Frame: as for outcome 1
Population: ITT population included all participants who were randomized to study treatment under PV >=5.0, regardless of whether or not they received study treatment. Here, "N" signifies number of participants evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Selinexor 60 mg (PV >=5) (Equivalent to 35 mg/m^2) | Physician's Choice 2 (PV >=5)
Number analyzed (Participants) | 14 | 2
Days | 175.0 [61.0 to 288.0] | 106.0 [NA to NA] — Upper and lower limits of 95% CI was not estimable due to the small number of participants and events.

7. Secondary Outcome: Percentage of Participants With Overall Response Rate (ORR)
Description: Overall response rate was defined as the point estimate of the percentage of participants who achieved CR (disappearance of all target and non-target lesions), partial response (PR) (>=30 % decrease in sum of longest diameters of target lesions taking as reference baseline sum longest diameters associated to non-progressive disease response for non-target lesions). CRi; < 5% BM blasts with residual neutropenia [ANC < 1000 cells/microL] or thrombocytopenia [platelets < 100,000/microL]. CRp; All criteria for CR except for residual neutropenia (<1x10^9/L) or thrombocytopenia (<100 x10^9/L) and morphologic leukemia-free state (MLFS); morphologic BM blast clearance to <5% in a marrow sample in which <=200 cells enumerated or cellularity is ≥10%, in absence of blasts with Auer rods, no hematologic recovery required.
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Selinexor 60 mg (PV >=5) (Equivalent to 35 mg/m^2) | Physician's Choice 2 (PV >=5)
Number analyzed (Participants) | 118 | 57
Percentage of participants | 13.6 [8.0 to 21.1] | 8.8 [2.9 to 19.3]

8. Secondary Outcome: Duration of Response (DOR)
Description: DOR was calculated from date of response of CR, CRi, CRp, MLFS, or PR to date of progression or recurrence based on IWG criteria. CR: <5% myeloblasts in bone marrow,absence of circulating blasts, hematologic recovery (peripheral blood ANC >1000 cells/microL, platelet count > 100,000/microL, no need for RBC transfusions), absence of extramedullary disease. PR: No circulating blasts, neutrophil count > =1.0 x10^9/L, platelet count >= 100 x10^9/L, >= 50 % reduction in bone marrow blast to 6% to 25%, or blasts less than or equal to (<=) 5% if Auer rods are present. CRp: All criteria for CR except for residual neutropenia (<1x10^9/L) or thrombocytopenia (<100 x10^9/L), CRi; < 5% bone marrow blasts with residual neutropenia [ANC < 1000 cells/microL] or thrombocytopenia [platelets < 100,000/microL]. MLFS: morphologic bone marrow blast clearance to < 5% in marrow sample, <= 200 cells enumerated/cellularity is ≥ 10%, in absence of blasts with Auer rods, no hematologic recovery required.
Time Frame: as for outcome 1
Population: ITT population included all participants who were randomized to study treatment under PV>=5.0, regardless of whether or not they received study treatment. Here, "N" signifies number of participants evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Selinexor 60 mg (PV >=5) (Equivalent to 35 mg/m^2) | Physician's Choice 2 (PV >=5)
Number analyzed (Participants) | 16 | 5
Days | 204.0 [117.0 to 334.0] | 148.0 [85.0 to NA] — Upper limit of 95% CI was not estimated due to less number of participants and events.

9. Secondary Outcome: Percentage of Participants With Disease Control Rate (DCR)
Description: DCR:Point estimate of % of participants with CR,CRi,CRp,MLFS,PR, or SD for <=4 weeks.CR:<5% myeloblasts in bone marrow (BM),absence of circulating blasts,hematologic recovery(peripheral blood ANC >1000 cells/microL and platelet count >100,000/microL, no need of RBC transfusions),absence of extramedullary disease. PR:No circulating blasts,Neutrophil count >=1.0 x10^9/L, Platelet count >= 100*10^9/L, >=50% reduction in BM blast to 6% to 25%, or blasts <=5% if Auer rods are present.CRp:All criteria for CR except for residual neutropenia (<1*10^9/L) or thrombocytopenia(<100 x10^9/L),CRi;< 5% BM blasts with residual neutropenia [ANC < 1000 cells/microL] or thrombocytopenia [platelets < 100,000/microL]. MLFS:morphologic BM blast clearance to <5% in a marrow sample in which <=200 cells enumerated or cellularity is ≥10%,in absence of blasts with Auer rods,no hematologic recovery required,SD:failure to achieve a response but not meeting criteria for disease progression over period of >4 weeks.
Time Frame: Up to 4 weeks from the date of randomization to the date of progression or recurrence based on IWG criteria
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Selinexor 60 mg (PV >=5) (Equivalent to 35 mg/m^2) | Physician's Choice 2 (PV >=5)
Number analyzed (Participants) | 118 | 57
Percentage of participants | 50.8 [41.5 to 60.2] | 40.4 [27.6 to 54.2]

10. Secondary Outcome: Duration of Disease Control Rate
Description: Duration of DCR calculated for all participants with DCR. CR: < 5% myeloblasts in BM, absence of circulating blasts, hematologic recovery (peripheral blood ANC >1000 cells/microL and platelet count > 100,000/microL, no need for RBC transfusions), absence of extra medullary disease. PR: No circulating blasts, Neutrophil count >=1.0 x 10^9/L, Platelet count >= 100 x 10^9/L, >= 50 % reduction in BM blast to 6% to 25%, or blasts <= 5% if Auer rods are present. CRp: All criteria for CR except for residual neutropenia (<1 x 10^9/L) or thrombocytopenia (<100 x 10^9/L), CRi; < 5% BM blasts with residual neutropenia [ANC < 1000 cells/microL] or thrombocytopenia [platelets < 100,000/microL]. MLFS; morphologic BM blast clearance to < 5% in a marrow sample in which <=200 cells enumerated/cellularity is >= 10%, in absence of blasts with Auer rods, no hematologic recovery required and SD; failure to achieve a response but not meeting criteria for disease progression over period of > 4 weeks.
Time Frame: Up to 4 weeks from the date of randomization to the date of progression or recurrence based on IWG criteria
Population: ITT population included all participants who were randomized to study treatment under PV>=5.0, regardless of whether or not they received study treatment. Here," N" signifies number of participants evaluable for this measure.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Selinexor 60 mg (PV >=5) (Equivalent to 35 mg/m^2) | Physician's Choice 2 (PV >=5)
Number analyzed (Participants) | 60 | 23
Days | 187.0 [125.0 to 261.0] | 233.0 [155.0 to 263.0]

11. Secondary Outcome: Change From Baseline in Quality of Life (QoL) and Patient-Reported Outcomes (Functional Assessment of Cancer Therapy -Leukemia [FACT-Leu]
Description: QoL was assessed by the FACT-Leu. FACT-Leu combines the General version of the Functional Assessment of Cancer Therapy (FACT-G) with a leukemia-specific sub-scale (17 items). The sub-scales for the FACT-G are Physical Well-Being (7 items), Social/Family Well-Being (7 items), Emotional Well-Being (6 items), and Functional Well-Being (7 items). The trial outcomes index (TOI; total of 31 items) was the primary measurement of interest, comprising the Physical and Functional sub-scales plus the leukemia - specific sub-scale. Each item was rated on a 5-point Likert scale. Range from 0 = (Not at all) to 4 = (Very much); therefore, the TOI had a score ranging from 0 to 124. Higher scores indicated improvement in well being. The QoL assessment was performed at baseline (prior to first dose of study treatment), Day 1 of each cycle on or after the second, and at the final visit.
Time Frame: Baseline, Day 1 of each treatment cycle (a maximum of 20 cycles: 28 days per cycle) up to 30 days after last dose of study drug (final visit)
Population: Per-Protocol (PP) population: all participants randomized to study treatment under PV>=5.0 who received any amount of study treatment and had no major protocol violations that compromised assessment of efficacy. Here, N= number of participants evaluable for this measure and n=participants evaluable for this outcome measure at specified categories.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Selinexor 60 mg (PV >=5) (Equivalent to 35 mg/m^2) | Physician's Choice 2 (PV >=5)
Number analyzed (Participants) | 71 | 34
Units on a scale
  Baseline: number analyzed (Participants) | 65 | 29
  Baseline | 70.5 (15.20) | 75.4 (14.74)
  C2D1: number analyzed (Participants) | 59 | 25
  C2D1 | 0.5 (16.50) | -1.9 (15.18)
  C3D1: number analyzed (Participants) | 39 | 16
  C3D1 | -1.9 (16.88) | -5.4 (22.25)
  C4D1: number analyzed (Participants) | 26 | 7
  C4D1 | -1.2 (15.70) | -7.4 (25.41)
  C5D1: number analyzed (Participants) | 20 | 7
  C5D1 | -2.4 (16.84) | 1.9 (8.40)
  C6D1: number analyzed (Participants) | 19 | 6
  C6D1 | -3.4 (15.66) | -4.7 (13.20)
  C7D1: number analyzed (Participants) | 15 | 5
  C7D1 | -5.0 (17.21) | -11.8 (27.43)
  C8D1: number analyzed (Participants) | 15 | 5
  C8D1 | -3.9 (15.78) | -10.6 (7.83)
  C9D1: number analyzed (Participants) | 11 | 4
  C9D1 | -2.7 (7.47) | -8.0 (8.49)
  C10D1: number analyzed (Participants) | 9 | 3
  C10D1 | 2.4 (13.19) | -10.7 (12.70)
  C11D1: number analyzed (Participants) | 7 | 2
  C11D1 | -0.1 (8.65) | -10.0 (9.90)
  C12D1: number analyzed (Participants) | 6 | 2
  C12D1 | -3.7 (11.69) | -7.0 (16.97)
  C13D1: number analyzed (Participants) | 4 | 1
  C13D1 | -3.3 (6.40) | -9.0 (NA) — Standard Deviation was not estimated due to less number of participants.
  C14D1: number analyzed (Participants) | 3 | 1
  C14D1 | -4.0 (3.46) | -15.0
  C15D1: number analyzed (Participants) | 2 | 1
  C15D1 | 1.5 (3.54) | -10.0 (NA) — Standard Deviation was not estimated due to less number of participants.
  C16D1: number analyzed (Participants) | 0 | 1
  C16D1 |  | -15.0 (NA) — Standard Deviation was not estimated due to less number of participants.
  C17D1: number analyzed (Participants) | 1 | 1
  C17D1 | -15.0 (NA) — Standard Deviation was not estimated due to less number of participants. | -7.0 (NA) — Standard Deviation was not estimated due to less number of participants.
  C18D1: number analyzed (Participants) | 1 | 0
  C18D1 | -1.0 (NA) — Standard Deviation was not estimated due to less number of participants. |
  C19D1: number analyzed (Participants) | 1 | 0
  C19D1 | -12.0 (NA) — Standard Deviation was not estimated due to less number of participants. |
  C20D1: number analyzed (Participants) | 1 | 0
  C20D1 | -14.0 (NA) — Standard Deviation was not estimated due to less number of participants. |
  Final visit: number analyzed (Participants) | 25 | 12
  Final visit | 2.5 (17.71) | -1.7 (20.46)

12. Secondary Outcome: Change From Baseline in European Quality of Life-5 Dimension (EQ-5D) Health Questionnaire Visual Analogue Scale (VAS)
Description: EQ-5D descriptive system comprises of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: 1=no problems, 2=slight problems, 3=moderate problems, 4=severe problems, and 5=extreme problems. EQ-5D-5L is a standardized instrument that measures health-related quality of life for men with prostate cancer. EQ-5D consists of EQ-5D descriptive system and EQ VAS. EQ-5D-5-VAS records participant's self-rated health on a vertical VAS that allows them to indicate their health state that can range from 0 (worst imaginable) to 100 (best imaginable), higher scores indicating a better health state.
Time Frame: as for outcome 11
Population: PP Population included all participants randomized to study treatment under PV >=5.0 who received any amount of study treatment and who had no major protocol violations that compromised assessment of efficacy. Here, N= number of participants evaluable for this measure and n =Participants evaluable for this outcome measure at specified categories
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Selinexor 60 mg (PV >=5) (Equivalent to 35 mg/m^2) | Physician's Choice 2 (PV >=5)
Number analyzed (Participants) | 71 | 34
Units on a scale
  Baseline: number analyzed (Participants) | 59 | 30
  Baseline | 67.9 (19.51) | 63.5 (21.10)
  C2D1: number analyzed (Participants) | 51 | 25
  C2D1 | -7.5 (23.45) | 0.8 (15.82)
  C3D1: number analyzed (Participants) | 35 | 17
  C3D1 | -13.3 (25.04) | -5.2 (23.54)
  C4D1: number analyzed (Participants) | 23 | 9
  C4D1 | -6.1 (20.80) | -5.0 (11.46)
  C5D1: number analyzed (Participants) | 18 | 10
  C5D1 | -0.9 (20.83) | -2.0 (15.31)
  C6D1: number analyzed (Participants) | 17 | 7
  C6D1 | -11.2 (25.90) | -1.4 (24.10)
  C7D1: number analyzed (Participants) | 14 | 5
  C7D1 | -3.7 (23.91) | 4.0 (10.84)
  C8D1: number analyzed (Participants) | 13 | 5
  C8D1 | 0.1 (16.77) | 5.0 (9.35)
  C9D1: number analyzed (Participants) | 9 | 4
  C9D1 | 4.6 (13.25) | 5.0 (10.80)
  C10D1: number analyzed (Participants) | 7 | 4
  C10D1 | 0.7 (18.58) | 6.3 (15.48)
  C11D1: number analyzed (Participants) | 6 | 2
  C11D1 | 0.8 (18.55) | -5.0 (21.21)
  C12D1: number analyzed (Participants) | 6 | 2
  C12D1 | 3.3 (16.63) | -5.0 (28.28)
  C13D1: number analyzed (Participants) | 3 | 1
  C13D1 | 6.7 (20.21) | 10.0 (NA) — Standard Deviation was not estimated due to less number of participants.
  C14D1: number analyzed (Participants) | 3 | 1
  C14D1 | 6.7 (25.66) | 15.0 (NA) — Standard Deviation was not estimated due to less number of participants.
  C15D1: number analyzed (Participants) | 2 | 1
  C15D1 | 3.5 (30.41) | -10.0 (NA) — Standard Deviation was not estimated due to less number of participants.
  C16D1: number analyzed (Participants) | 0 | 1
  C16D1 |  | 20.0 (NA) — Standard Deviation was not estimated due to less number of participants.
  C17D1: number analyzed (Participants) | 1 | 1
  C17D1 | 25.0 (NA) — Standard Deviation was not estimated due to less number of participants. | -5.0 (NA) — Standard Deviation was not estimated due to less number of participants.
  C18D1: number analyzed (Participants) | 1 | 0
  C18D1 | 25.0 (NA) — Standard Deviation was not estimated due to less number of participants. |
  C19D1: number analyzed (Participants) | 1 | 0
  C19D1 | 30.0 (NA) — Standard Deviation was not estimated due to less number of participants. |
  C20D1: number analyzed (Participants) | 1 | 0
  C20D1 | 35.0 (NA) — Standard Deviation was not estimated due to less number of participants. |

ADVERSE EVENTS:
Time Frame: From start of study drug administration to 30 days after last dose of study drug (approximately 48 months)
Description: Same event may appear as both an adverse event (AE) and a serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study. AEs and SAEs were collected for safety population.
Groups:
- Selinexor Approximately 55 mg/m^2 (60 to 120 mg Based on BSA): Participants under PV <5.0 (those who had one prior line of AML therapy), received oral selinexor tablets at a dose of approximately 55 mg/m^2 (60 to 120 mg based on BSA) twice weekly, on Day 1 and 3 of each week of 4-week cycle (28 days per cycle).
- Selinexor 60mg (PV<5) (Equivalent to 35 mg/m^2): Participants under PV <5.0 (those who had one prior line of AML therapy), received oral selinexor tablets at a fixed dose of 60 mg (equivalent to 35 mg/m^2), based on BSA, twice weekly, on Day 1 and 3 of each week of 4-week cycle (28 days per cycle).
- Selinexor 60mg (PV >=5) (Equivalent to 35 mg/m^2): Participants under PV >=5 (PV 5: those who had at least one prior line of AML therapy, PV 5.1: who had at least two prior line of AML therapy), received oral selinexor tablets at a dose of 60 mg (equivalent to 35 mg/m^2) twice weekly, on Day 1 and 3 of each week of 4- week cycle (28 days per cycle).
Arm/Group | Selinexor Approximately 55 mg/m^2 (60 to 120 mg Based on BSA) | Selinexor 60mg (PV<5) (Equivalent to 35 mg/m^2) | Selinexor 60mg (PV >=5) (Equivalent to 35 mg/m^2) | Physician's Choice 1 (PV <5) | Physician's Choice 2 (PV >=5)
All-Cause Mortality (participants affected / at risk) | 24/71 | 3/27 | 28/115 | 7/39 | 9/45
Serious Adverse Events (participants affected / at risk) | 58/71 | 15/27 | 89/115 | 25/39 | 30/45
Other Adverse Events (participants affected / at risk) | 71/71 | 27/27 | 113/115 | 37/39 | 40/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Selinexor Approximately 55 mg/m^2 (60 to 120 mg Based on BSA) (N=71) | Selinexor 60mg (PV<5) (Equivalent to 35 mg/m^2) (N=27) | Selinexor 60mg (PV >=5) (Equivalent to 35 mg/m^2) (N=115) | Physician's Choice 1 (PV <5) (N=39) | Physician's Choice 2 (PV >=5) (N=45)
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 2 | 0 | 3
Febrile Neutropenia (Blood and lymphatic system disorders) | 16 | 4 | 20 | 8 | 16
Leukostasis Syndrome (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 0
Splenic Infarction (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 1 | 0 | 0
Acute Coronary Syndrome (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 2 | 0 | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Cardiac Failure (Cardiac disorders) | 1 | 0 | 3 | 0 | 0
Cardiac Failure Congestive (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Cardio-Respiratory Arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Sinus Bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Tachyarrhythmia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Ventricular Fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 3 | 0 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 6 | 0 | 0
Diverticular Perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0
Large Intestinal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Mouth Ulceration (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Tooth Loss (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 4 | 0 | 3 | 0 | 0
Asthenia (General disorders) | 3 | 0 | 2 | 2 | 0
Condition Aggravated (General disorders) | 0 | 0 | 0 | 0 | 1
General Physical Health Deterioration (General disorders) | 1 | 0 | 2 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 1 | 0
Multiple Organ Dysfunction Syndrome (General disorders) | 1 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 4 | 1 | 7 | 2 | 1
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 0 | 2 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Arthritis Bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Aspergillus Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Biliary Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Biliary Tract Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 2 | 0 | 1 | 1 | 1
Clostridium Difficile Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Device Related Infection (Infections and infestations) | 0 | 0 | 1 | 1 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Escherichia Sepsis (Infections and infestations) | 1 | 0 | 0 | 1 | 1
Fungal Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 2
Klebsiella Sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Lung Infection (Infections and infestations) | 3 | 1 | 1 | 3 | 0
Necrotising Fasciitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Neutropenic Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Penile Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Perirectal Abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pneumocystis Jirovecii Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 10 | 4 | 10 | 4 | 3
Pneumonia Fungal (Infections and infestations) | 2 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 8 | 1 | 3 | 3 | 1
Septic Shock (Infections and infestations) | 1 | 0 | 3 | 1 | 0
Sialoadenitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Skin Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Soft Tissue Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 3 | 1 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Vaginal Abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Vulval Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 1
Femur Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Subarachnoid Haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Subdural Haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0
Subdural Haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Blood Alkaline Phosphatase Increased (Investigations) | 1 | 0 | 0 | 0 | 0
C-Reactive Protein Increased (Investigations) | 0 | 0 | 1 | 0 | 0
Electrocardiogram Change (Investigations) | 0 | 0 | 1 | 0 | 0
Enterococcus Test Positive (Investigations) | 0 | 0 | 0 | 1 | 0
Troponin T Increased (Investigations) | 0 | 0 | 1 | 0 | 0
Vitamin B12 Decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Weight Decreased (Investigations) | 1 | 0 | 1 | 0 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 0 | 6 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 5 | 0 | 2 | 1 | 0
Failure To Thrive (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Fluid Overload (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0
Hypercreatininaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 1 | 0 | 0 | 0
Hypophagia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Cerebellar Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Cerebral Haemorrhage (Nervous system disorders) | 1 | 0 | 2 | 0 | 1
Cerebral Infarction (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Cerebrovascular Accident (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 2 | 0 | 0
Embolic Stroke (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Haemorrhage Intracranial (Nervous system disorders) | 2 | 0 | 1 | 0 | 0
Haemorrhagic Cerebral Infarction (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Ischaemic Stroke (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Loss Of Consciousness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Nervous System Disorders (Nervous system disorders) | 8 | 1 | 15 | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 2 | 1 | 3 | 0 | 0
Confusional State (Psychiatric disorders) | 4 | 0 | 2 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Mental Status Changes (Psychiatric disorders) | 1 | 0 | 2 | 0 | 0
Organic Brain Syndrome (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Acute Kidney Injury (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Oliguria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Renal Failure (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Vaginal Haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pulmonary Mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2 | 0 | 0
Social Stay Hospitalisation (Social circumstances) | 0 | 1 | 0 | 0 | 0
Aortic Aneurysm (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 4 | 0 | 0
Peripheral Ischaemia (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Thrombophlebitis (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Venous Thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 8 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Selinexor Approximately 55 mg/m^2 (60 to 120 mg Based on BSA) (N=71) | Selinexor 60mg (PV<5) (Equivalent to 35 mg/m^2) (N=27) | Selinexor 60mg (PV >=5) (Equivalent to 35 mg/m^2) (N=115) | Physician's Choice 1 (PV <5) (N=39) | Physician's Choice 2 (PV >=5) (N=45)
Nausea (Gastrointestinal disorders) | 41 (41) | 16 (16) | 68 (68) | 13 (13) | 8 (8)
Diarrhoea (Gastrointestinal disorders) | 17 (17) | 13 (13) | 41 (41) | 8 (8) | 6 (6)
Constipation (Gastrointestinal disorders) | 20 (20) | 8 (8) | 25 (25) | 16 (16) | 15 (15)
Vomiting (Gastrointestinal disorders) | 19 (19) | 10 (10) | 30 (30) | 7 (7) | 6 (6)
Stomatitis (Gastrointestinal disorders) | 8 (8) | 0 (0) | 8 (8) | 3 (3) | 3 (3)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 12 (12) | 2 (2) | 6 (6)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 6 (6) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 2 (2) | 3 (3) | 1 (1) | 1 (1)
Gingival Bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 7 (7) | 1 (1) | 2 (2)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 3 (3)
Aphthous Ulcer (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 2 (2)
Mouth Haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 4 (4) | 1 (1) | 0 (0)
Abdominal Discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 2 (2)
Gingival Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Toothache (Gastrointestinal disorders) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Dry Mouth (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Oral Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Abdominal Pain Lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anal Fissure (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Angina Bullosa Haemorrhagica (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Eructation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mouth Ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Oral Disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Oral Mucosa Haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Oral Mucosal Blistering (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal Tenderness (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal Incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breath Odour (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Faeces Soft (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gingival Hypertrophy (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Glossitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inguinal Hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lip Blister (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip Dry (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lip Oedema (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lip Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lip Swelling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lip Ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mouth Swelling (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral Contusion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral Dysaesthesia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palatal Disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Perianal Erythema (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rectal Fissure (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retching (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Salivary Hypersecretion (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tongue Haematoma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tongue Ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth Loss (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Trichoglossia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 33 (33) | 13 (13) | 50 (50) | 15 (15) | 13 (13)
Pyrexia (General disorders) | 8 (8) | 5 (5) | 28 (28) | 13 (13) | 13 (13)
Oedema Peripheral (General disorders) | 17 (17) | 5 (5) | 21 (21) | 10 (10) | 5 (5)
Asthenia (General disorders) | 17 (17) | 6 (6) | 22 (22) | 5 (5) | 5 (5)
Malaise (General disorders) | 2 (2) | 1 (1) | 8 (8) | 3 (3) | 1 (1)
Oedema (General disorders) | 2 (2) | 0 (0) | 5 (5) | 4 (4) | 2 (2)
Chills (General disorders) | 1 (1) | 1 (1) | 5 (5) | 3 (3) | 1 (1)
Mucosal Inflammation (General disorders) | 3 (3) | 0 (0) | 1 (1) | 4 (4) | 3 (3)
Pain (General disorders) | 0 (0) | 0 (0) | 7 (7) | 1 (1) | 1 (1)
Gait Disturbance (General disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
General Physical Health Deterioration (General disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Injection Site Bruising (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Non-Cardiac Chest Pain (General disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Ulcer (General disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Catheter Site Haemorrhage (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Face Oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Generalised Oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Secretion Discharge (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Catheter Site Haematoma (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug Intolerance (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Extravasation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling Cold (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Granuloma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hernia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Impaired Healing (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion Site Haemorrhage (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection Site Discolouration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection Site Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mucosal Dryness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nodule (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral Swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased Appetite (General disorders) | 41 (41) | 12 (12) | 61 (61) | 9 (9) | 7 (7)
Hyponatraemia (Metabolism and nutrition disorders) | 26 (26) | 6 (6) | 25 (25) | 3 (3) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 10 (10) | 1 (1) | 9 (9) | 5 (5) | 6 (6)
Hypocalcaemia (Metabolism and nutrition disorders) | 5 (5) | 2 (2) | 11 (11) | 2 (2) | 4 (4)
Hypercreatininaemia (Metabolism and nutrition disorders) | 5 (5) | 0 (0) | 13 (13) | 2 (2) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 7 (7) | 0 (0) | 9 (9) | 2 (2) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 6 (6) | 3 (3) | 7 (7) | 1 (1) | 3 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 8 (8) | 2 (2) | 9 (9) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 8 (8) | 0 (0) | 6 (6) | 3 (3) | 2 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 9 (9) | 1 (1) | 5 (5) | 0 (0) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 5 (5) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 (4) | 1 (1) | 1 (1) | 2 (2) | 2 (2)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0)
Hypermagnesaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Hyperlipasaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fluid Retention (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyperamylasaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Fluid Overload (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour Lysis Syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Failure To Thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemic Hyperosmolar Nonketotic Syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhomocysteinaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypouricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metabolic Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Polydipsia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 29 (29) | 7 (7) | 38 (38) | 18 (18) | 11 (11)
Anaemia (Blood and lymphatic system disorders) | 20 (20) | 7 (7) | 29 (29) | 17 (17) | 10 (10)
Neutropenia (Blood and lymphatic system disorders) | 6 (6) | 5 (5) | 17 (17) | 10 (10) | 9 (9)
Leukopenia (Blood and lymphatic system disorders) | 2 (2) | 3 (3) | 10 (10) | 5 (5) | 4 (4)
Febrile Neutropenia (Blood and lymphatic system disorders) | 9 (9) | 2 (2) | 7 (7) | 3 (3) | 2 (2)
Leukocytosis (Blood and lymphatic system disorders) | 6 (6) | 2 (2) | 6 (6) | 4 (4) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Increased Tendency To Bruise (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Polycythaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Splenomegaly (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14 (14) | 5 (5) | 24 (24) | 8 (8) | 10 (10)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 3 (3) | 25 (25) | 7 (7) | 7 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 3 (3) | 15 (15) | 5 (5) | 8 (8)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 3 (3) | 2 (2) | 3 (3)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 3 | 3 (3) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 4 (4) | 1 (1) | 1 (1)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 4 (4) | 0 (0) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper-Airway Cough Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung Consolidation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung Infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal Dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal Inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paranasal Sinus Discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngeal Inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary Mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rales (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus Disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tonsillar Erythema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tonsillar Hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 6 (6) | 2 (2) | 9 (9) | 5 (5) | 2 (2)
Oral Herpes (Infections and infestations) | 2 (2) | 0 (0) | 3 (3) | 4 (4) | 4 (4)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 5 (5) | 1 (1) | 3 (3)
Oral Candidiasis (Infections and infestations) | 4 (4) | 0 (0) | 4 (4) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 4 (4) | 3 (3) | 1 (1)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Lung Infection (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Device Related Infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Periodontitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Pneumonia Fungal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Sepsis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Candida Infection (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Oesophageal Candidiasis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Skin Infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Staphylococcal Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Clostridium Difficile Colitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Clostridium Difficile Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Ear Infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fungal Infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Herpes Dermatitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lip Infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nasal Herpes (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pseudomonas Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rash Pustular (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Rhinovirus Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Soft Tissue Infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess Limb (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anal Abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspergillus Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asymptomatic Bacteriuria (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacterial Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bacteriuria (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter Site Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Clostridium Colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermo-Hypodermitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Empyema (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Encephalitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterobiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Enterococcal Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Genital Herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Groin Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes Simplex (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes Zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infected Dermal Cyst (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymph Gland Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meningitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metapneumovirus Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucosal Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oesophageal Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ophthalmic Herpes Simplex (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral Fungal Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Parotitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia Klebsiella (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proteus Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pseudomembranous Colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Septic Shock (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sialoadenitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal Bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stenotrophomonas Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tonsillitis Bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth Abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Varicella Zoster Virus Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 7 (7) | 3 (3) | 12 (12) | 3 (3) | 2 (2)
Headache (Nervous system disorders) | 5 (5) | 3 (3) | 3 (3) | 7 (7) | 6 (6)
Syncope (Nervous system disorders) | 3 (3) | 1 (1) | 5 (5) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 12 (12) | 2 (2) | 18 (18) | 8 (8) | 2 (2)
Presyncope (Nervous system disorders) | 1 (1) | 3 (3) | 3 (3) | 0 (0) | 2 (2)
Somnolence (Nervous system disorders) | 4 (4) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Ageusia (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Balance Disorder (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Memory Impairment (Nervous system disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cognitive Disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dysarthria (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy Peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Speech Disorder (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aphonia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cogwheel Rigidity (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coordination Abnormal (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drooling (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhage Intracranial (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemianopia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hemianopia Homonymous (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypersomnia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyposmia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Parosmia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sensory Loss (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Synaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight Decreased (Investigations) | 15 (15) | 4 (4) | 20 (20) | 3 (3) | 3 (3)
Alanine Aminotransferase Increased (Investigations) | 2 (2) | 2 (2) | 5 (5) | 2 (2) | 1 (1)
Aspartate Aminotransferase Increased (Investigations) | 2 (2) | 0 (0) | 5 (5) | 2 (2) | 1 (1)
International Normalised Ratio Increased (Investigations) | 1 (1) | 2 (2) | 4 (4) | 3 (3) | 0 (0)
Weight Increased (Investigations) | 2 (2) | 1 (1) | 0 (0) | 6 (6) | 1 (1)
Blood Lactate Dehydrogenase Increased (Investigations) | 5 (5) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Blood Alkaline Phosphatase Increased (Investigations) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
C-Reactive Protein Increased (Investigations) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Blood Uric Acid Increased (Investigations) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Electrocardiogram Qt Prolonged (Investigations) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Activated Partial Thromboplastin Time Prolonged (Investigations) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Blood Creatine Phosphokinase Increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Blood Thyroid Stimulating Hormone Increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
General Physical Condition Abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Blood Creatine Phosphokinase Decreased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood Pressure Decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blood Urea Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cardiac Murmur (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Ejection Fraction Decreased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram Change (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypophonesis (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Oxygen Saturation Decreased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Transaminases Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alpha 1 Foetoprotein Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Astrovirus Test Positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bilirubin Urine (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blast Cell Count Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bleeding Time Prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood Alkaline Phosphatase Decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood Lactic Acid Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood Test Abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Body Temperature Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gamma-Glutamyltransferase Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Glomerular Filtration Rate Decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Liver Function Test Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prothrombin Time Prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White Blood Cell Count (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White Blood Cell Count Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Night Sweats (Skin and subcutaneous tissue disorders) | 8 (8) | 3 (3) | 10 (10) | 1 (1) | 4 (4)
Petechiae (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0) | 3 (3) | 7 (7) | 6 (6)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 6 (6) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 4 (4) | 2 (2)
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 2 (2)
Ecchymosis (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
Skin Lesion (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Cold Sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Skin Mass (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Swelling Face (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermal Cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis Bullous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Facial Wasting (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Macule (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nail Disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Photosensitivity Reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash Erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash Pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin Discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin Induration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin Maceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 10 (10) | 4 (4) | 7 (7) | 4 (4) | 3 (3)
Confusional State (Psychiatric disorders) | 5 (5) | 2 (2) | 8 (8) | 2 (2) | 3 (3)
Anxiety (Psychiatric disorders) | 2 (2) | 2 (2) | 4 (4) | 2 (2) | 1 (1)
Depression (Psychiatric disorders) | 2 (2) | 2 (2) | 2 (2) | 3 (3) | 1 (1)
Agitation (Psychiatric disorders) | 6 (6) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hallucination (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Personality Change (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Abnormal Dreams (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bulimia Nervosa (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Disorientation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flat Affect (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hallucination, Visual (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Irritability (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Listless (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental Disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental Status Changes (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nervousness (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Psychomotor Retardation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 0 (0) | 6 (6) | 5 (5) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 6 (6) | 5 (5) | 5 (5)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 5 (5) | 0 (0) | 4 (4) | 3 (3) | 0 (0)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 3 (3) | 1 (1) | 2 (2)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 3 (3)
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 5 (5) | 1 (1) | 0 (0)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypercreatinaemia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint Swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pain In Jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Groin Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ligament Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Limb Discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb Mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle Mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle Tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle Twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Torticollis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 6 (6) | 1 (1) | 11 (11) | 4 (4) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 2 (2) | 5 (5) | 7 (7) | 1 (1)
Hypertension (Vascular disorders) | 4 (4) | 2 (2) | 2 (2) | 1 (1) | 1 (1)
Pallor (Vascular disorders) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 1 (1)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Thrombophlebitis (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Orthostatic Hypotension (Vascular disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Circulatory Collapse (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot Flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intermittent Claudication (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Poor Peripheral Circulation (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombophlebitis Superficial (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Venous Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 8 (8) | 2 (2) | 3 (3) | 2 (2) | 3 (3)
Haematuria (Renal and urinary disorders) | 3 (3) | 3 (3) | 1 (1) | 2 (2) | 3 (3)
Pollakiuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 3 (3) | 1 (1) | 2 (2)
Proteinuria (Renal and urinary disorders) | 3 (3) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Renal Failure (Renal and urinary disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Urinary Incontinence (Renal and urinary disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Bladder Dilatation (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic Kidney Disease (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Micturition Urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bladder Pain (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chromaturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nocturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Polyuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urethral Caruncle (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urethral Haemorrhage (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urge Incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary Tract Obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary Tract Pain (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vision Blurred (Eye disorders) | 8 (8) | 1 (1) | 9 (9) | 1 (1) | 0 (0)
Visual Impairment (Eye disorders) | 4 (4) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Dry Eye (Eye disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Visual Acuity Reduced (Eye disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Conjunctival Haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Eye Pain (Eye disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Lacrimation Increased (Eye disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Eye Haemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eyelid Oedema (Eye disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Ocular Hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Periorbital Oedema (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Photopsia (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal Haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye Inflammation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye Swelling (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eyelid Ptosis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitreous Floaters (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vitreous Haemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 6 (6) | 2 (2) | 9 (9) | 2 (2) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 5 (5) | 2 (2) | 5 (5) | 3 (3) | 1 (1)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Procedural Pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Skin Abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transfusion Reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Allergic Transfusion Reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Animal Bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Facial Bones Fracture (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Head Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Periorbital Haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post Procedural Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 5 (5) | 1 (1) | 4 (4) | 0 (0) | 2 (2)
Sinus Tachycardia (Cardiac disorders) | 4 (4) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Acute Left Ventricular Failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angina Pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bundle Branch Block Right (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac Failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac Flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Supraventricular Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia Paroxysmal (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deafness (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Ear Discomfort (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Ear Pain (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear Congestion (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eustachian Tube Dysfunction (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Excessive Cerumen Production (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 (2) | 0 (0) | 5 (5) | 1 (1) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatomegaly (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Jaundice (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ocular Icterus (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 4 (4) | 1 (1) | 0 (0)
Cushingoid (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast Pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast Swelling (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gynaecomastia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nipple Pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema Genital (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ovarian Cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Testicular Oedema (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaginal Haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute Myeloid Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chloroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukaemic Infiltration (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2015-08-04): https://cdn.clinicaltrials.gov/large-docs/41/NCT02088541/Prot_000.pdf
  • Statistical Analysis Plan (2016-09-30): https://cdn.clinicaltrials.gov/large-docs/41/NCT02088541/SAP_001.pdf